CLINICAL TRIAL: NCT02476305
Title: Evaluation of the Cryodestruction of Non Abdominopelvic Desmoid Tumors in Patients Progressing Despite Medical
Brief Title: Evaluation of the Cryodestruction of Non Abdominopelvic Desmoid Tumors in Patients Progressing Despite Medical Treatment
Acronym: CRYODESMO01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6018
Record Dates: First submitted 2015-06-04; First posted 2015-06-19 (Estimated); Last update posted 2026-01-20 (Actual); Status verified 2017-11

CONDITIONS: Desmoid Tumors
MeSH Terms: conditions — Desmoid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cryoablation (Experimental): patients undergo cryoablation procedure for desmoid tumor
  Interventions: Device: "cryoprobes"

INTERVENTIONS:
Device: "cryoprobes" — Patient undergo percutaneous cryoablation of desmoid tumor, with cryoprobes

SUMMARY:
Desmoid tumors (DT) are rare tumors (2-4 cases/million/year) that originate from musculoaponeurotic structures. Although they are benign tumors with no metastatic potential, DT are considered as locally aggressive tumors, with local invasiveness and tissue destruction, leading to pain, and disability. Surgery remains the keystone of therapy, but is limited by the anatomical situation of extra-abdominal desmoid (EAD) tumors (chest wall, root members). In patients where surgery is considered, negative-margin resection (R0) is recommended, but this frequently results in cosmetic/functional impairment. Moreover, prognostic impact of R0 resections remains controversial. The outcome after initial surgery depends upon several factors such as age, tumor site, and tumor size as demonstrated by recent data from the French Sarcoma Group.

Alternative therapies to DT surgery for front-line or recurrence include NSAID's, anti-estrogens alone or in combination, -interferon, chemotherapy, targeted therapies or radiation therapy. All of these medical approaches however may fail to achieve long-term disease control and a number of patients suffer from irreducible pain, and disability from tumor volume.

Cryoablation is a promising technique that is suitable for patients experiencing extra-abdominal DT. The procedure is based on repeated cycles of freezing/passive thawing of the tumor, leading to cell death. The technique has many advantages, among which: the accurate control of iceball under real-time MRI or CT-scan monitoring (that is not possible with other techniques such as radiofrequency), the lack of mutilation, the possibility of repeating the procedure. The cryoablation procedure has proven to be beneficial for the treatment of various tumors (liver metastases, breast, kidney). Recently, percutaneous cryotherapy has been reported in the treatment of EAD tumors poorly suited to surgery, with promising results.

In the light of these encouraging data, it is believed that patients with extra-abdominal DT not amenable to surgery unless unacceptable surgical sequel and progressing after at least two lines of adequate medical therapy (tamoxifen, NSAID or chemotherapy), could benefit from the cryoablation procedure. Tumor cryotherapy-induced regression should allow symptoms relief, prolonged progression-free survival and a better quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Extra-abdominal desmoid tumor (confirmed by prior biopsy)
* 18 years of age or older
* Tumor deemed accessible for cryoablation procedure by the operator in the investigator center
* At least one measurable lesion (RECIST v1.1) using MRI (gadolinium injection mandatory)
* 90 % of destruction of the tumor achievable in one procedure of cryoablation with a possible second cryoablation procedure (if a complete treatment must be achieved).
* Progressive disease under standard treatment (after at least two lines of adequate medical therapy, including tamoxifen, non-steroid anti-inflamatory or chemotherapy), with presence of functional symptoms and/or pain The definition of progressing tumors also involves patients with RECIST stable disease, but with persistent functional disability or tumor-induced pain not controlled by adequate pain medication including narcotics.
* Unresectable tumor or tumor amenable only to mutilating surgery, deemed inappropriate, and discussed in multidisciplinary meeting (RCP)
* ECOG performance status 0-2
* Biological and hematological parameters:

  * neutrophils 1,5.109/L
  * platelet count 100.109/L
  * No significant hemostatic abnormalities
* Subject affiliated to social security
* Signed informed consent

Exclusion Criteria:

* Any contra-indication for the procedure as stated by the radiologist in terms of tumor size, proximity to neural/vascular structures making the procedure at unacceptable risk
* Impaired hemostasis, that may interfere with the conduct of the cryoablation
* Concurrent participation in other experimental studies that could affect endpoints of this study
* Contraindication to any form of sedation
* Contraindication to MRI or gadolinium injection (proven allergy, subject with impaired renal function (defined by a creatinine clearance below 30 ml/min by MDRD formula))
* Psychiatric disorders and adults under guardianship
* Pregnancy or breastfeeding
* Patients under judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Non-progression of non-abdominopelvic desmoid tumor | 12 months
  The success of cryoablation, i.e. non-progression of non-abdominopelvic desmoid tumor, will be declared if the MRI control at 1 year after the last procedure shows:
  * no suspicious contrast enhancement (the suspicious character is defined by heterogeneous or nodular or crescent-shape contrast enhancement) in the treated zone,
  * and if the cryolesion (ablation zone) is not increasing in size compared to early post-ablation control (M1)

CONTACTS AND LOCATIONS:
Overall Officials: Afshin GANGI, MD, Principal Investigator — Strasbourg's University Hospitals
Locations (1):
- Service d'Imagerie Interventionnelle, Strasbourg, Alsace, France

REFERENCES:
- [Result] Kurtz JE, Buy X, Deschamps F, Sauleau E, Bouhamama A, Toulmonde M, Honore C, Bertucci F, Brahmi M, Chevreau C, Duffaud F, Gantzer J, Garnon J, Blay JY, Gangi A. CRYODESMO-O1: A prospective, open phase II study of cryoablation in desmoid tumour patients progressing after medical treatment. Eur J Cancer. 2021 Jan;143:78-87. doi: 10.1016/j.ejca.2020.10.035. Epub 2020 Dec 5. PMID 33290994